CLINICAL TRIAL: NCT06419907
Title: A Feasibility Study Evaluating the Impact of Differing Completion Rates of a Face-to-face Diabetes Self-management Education Programme on Patient Reported Outcome Measures.
Brief Title: Differing Completion Rates of DIABETES Education on Patient Reported Outcomes
Acronym: DIABETES-PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: St Helens & Knowsley Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UoL001848; 337691 (Other: IRAS)
Record Dates: First submitted 2024-05-09; First posted 2024-05-17 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus, Type 2; Patient Education as Topic
Keywords: health education; patient reported outcome measures; type 2 diabetes mellitus; patient education as topic
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Active Comparator): 100% of a face to face 6 hour structured diabetes self management education session
  Interventions: Behavioral: Type 2 Live Well (structured diabetes self management education programme)
- Group 2 (Experimental): 60% of a face to face 6 hour structured diabetes self management education session. Total attendance will be 3 hours 36 minutes.
  Interventions: Behavioral: Type 2 Live Well (structured diabetes self management education programme)
- Group 3 (Experimental): 10% of a face to face 6 hour structured diabetes self management education session. Total attendance will be 36 minutes.
  Interventions: Behavioral: Type 2 Live Well (structured diabetes self management education programme)
- Group 4 (Active Comparator): Will not attend a face to face 6 hour structured diabetes self management education session
  Interventions: Behavioral: Type 2 Live Well (structured diabetes self management education programme)

INTERVENTIONS:
Behavioral: Type 2 Live Well (structured diabetes self management education programme) — Structured diabetes self management education programme designed to support those with type 2 diabetes self care and prevent long term associated complications.

SUMMARY:
The goal of this clinical feasibility trial is to test the impact of differing completion rates of a face-to-face diabetes self-management education programme on patient-reported outcomes measuring self-care, diabetes distress and quality of life in people with type 2 diabetes. The main question it aims to answer is:

1. What is the impact of differing completion rates of DSME programmes on ability to self-care (primary outcome), diabetes distress and health related quality of life in type 2 diabetes.

Researchers will compare participants across four study groups (Group 1 will receive a full DSME programme, Group 2 will receive 60%, Group 3 will receive 10% and Group 4 will have delayed education) to see if patients who attend minimal aspects (10%) of diabetes self-management education programmes gain clinically significant improvements in ability to self-care compared to those who do not attend and if the nationally accepted 60 % completion rate is as effective as 100% completion.

Participants will:

* complete three validated patient reported outcome measures testing self care activities, diabetes distress and health related quality of life.
* Attend structured diabetes self-management education of differing completion rates dependent on the group they have been allocated to.
* repeat the same three patient reported outcome measures 2-4 months after intervention. For participants in group 4 this will be 3-4 months from baseline.

DETAILED DESCRIPTION:
Structured diabetes self-management education (DSME) is internationally recommended for all people with newly diagnosed type 2 diabetes and is designed to support patients in self-managing their condition and prevent associated long-term complications. DSME is proven to be as effective as pharmacotherapy in preventing diabetes associated morbidity and premature mortality but attendance at both a national and local level remains poor. Local records suggest that of those that start DSME (9%) only 12.6% complete the programme. Attendance at DSME is currently benchmarked as having completed a registration form and had at least one active engagement with a programmes content, with 'completion' measured against ≥60% completion despite landmark trials reporting outcomes based on the full completion of a programme. Little is known, of the effectiveness of DSME on the psychological and emotional health of people with diabetes who complete less than the full DSME programme.

This feasibility study will test the impact of differing completion rates of a face-to-face DSME programme on patient reported outcomes measuring self-care, diabetes distress and quality of life in people with type 2 diabetes.

Using a quantitative approach, a single centre, randomised feasibility study will be conducted, aiming to recruit 120 eligible people with type 2 diabetes due to attend a secondary care diabetes clinic in the Northwest UK for specialist support, education and advice. Participants will be randomised into one of four groups: Group 1 will receive a full DSME programme, Group 2 will receive 60%, Group 3 will receive 10% and Group 4 will have delayed education. Normal clinical care will continue. Preliminary outcomes (psychometric questionnaire scores measuring ability to self-care, diabetes distress and health related quality of life) will be evaluated at baseline and 3-4 months post-intervention. Measures of feasibility (eligibility, recruitment and retention rates) will be reported.

Whilst the current literature evidences the clear benefits for people with type 2 diabetes attending DSME programmes, there is minimal understanding of the benefits of partial DSME completion on a person's ability to self-care despite national consensus accepting 60% attendance as 'completed'. The proposed research aims to test the feasibility of conducting a full randomised control trial to evaluate the effectiveness of DSME programmes on psychometric outcomes with differing completion rates

ELIGIBILITY:
Inclusion Criteria:

* All patients with a diagnosis of type 2 diabetes aged ≥18 years of age referred to the Diabetes centre who are able to provide informed consent and are responsible for daily management of their diabetes will be screened for entry into the study

Exclusion Criteria:

The following patients will be excluded entry into the study:

* Lack capacity to make an informed decision.
* A diagnosis of type 1, type 3c, Maturity-onset diabetes of the young (MODY) or gestational diabetes.
* Received structured education for their diabetes within the last 12 months either online or face to face.
* Require 1:1 education support e.g., requires interpreter.
* Patients unable to attend for structured classroom education e.g., housebound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gemma A Lewis, Principal Investigator — University of Liverpool
Locations (1):
- Diabetes Centre, St Helens Hospital, St Helens, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All metadata records for the qualitative data will be uploaded onto the University research data repository. All records will be anonymised and identified by study number only in order to maintain confidentiality.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available following the end of study and completion of associated publications and PhD thesis submission.

REFERENCES:
- [Derived] Lewis G, Irving G, Wilding J, Hardy K. Evaluating the impact of differing completion rates of a face-to-face DIABETES self-management education programme on Patient Reported Outcome measures (DIABETES PRO): A feasibility trial protocol. Diabet Med. 2024 Dec;41(12):e15430. doi: 10.1111/dme.15430. Epub 2024 Sep 5. PMID 39235931
- See also: Secure online environment for University of Liverpool Researchers to deposit, share and promote data and information — https://datacat.liverpool.ac.uk/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 120 participants consented and were randomised between May 2024 and February 2025 (30 per group). 68% of these were from secondary care clinics, 32% from primary care services (GP referrals and shared care reports).
Pre-assignment Details: Patients with a recorded clinical diagnosis of type 2 diabetes aged ≥18 years who met local and national eligibility criteria for DSME who could provide written informed consent and were responsible for daily management of their diabetes.
  Exclusion criteria include:
  * Lack capacity to make an informed decision.
  * Type 1, type 3c, monogenic or gestational diabetes.
  * Received structured education for diabetes within last 12 months either online or face to face.
  * Require 1:1 education
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 30 | 30 | 30 | 30
Completed | 30 | 27 | 28 | 28
Not Completed | 0 | 3 | 2 | 2
Not completed — Protocol Violation | 0 | 3 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Adherence was assessed during the study by reviewing the number of dropouts during the study and non-adherence to the randomised intervention. Four participants were not included in the final analysis due to protocol deviations: three attended structured education during the trial to meet their medical needs, one of whom was of mixed ethnicity, and another completed 100% DSME instead of the randomised 60%. A further 3 were lost to follow up.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 30 | 27 | 28 | 28 | 113
Age, Continuous [Median (Standard Deviation); unit: year] | 60 (13) | 62 (12) | 62 (17) | 60 (16) | 61 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 9 | 16 | 56
  Male | 13 | 13 | 19 | 12 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 27 | 28 | 28 | 113
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Index of multiple deprivation (IMD) [Median (Standard Deviation); unit: units on a scale] — The Indices of Multiple Deprivation (IMD) assigns a decile score to small areas (postcodes), ranking them from most to least deprived. Deciles are created by dividing all areas into ten equal groups based on their deprivation score, with decile 1 representing the most deprived 10% of areas and decile 10 representing the least deprived 10%. This allows for a relative comparison of deprivation levels across different patient postcodes.
  units on a scale | 3 (5) | 3 (4) | 2 (4) | 3 (4) | 3 (4)
Charlson Comorbidity index [Median (Standard Deviation); unit: units on a scale] — The Charlson Comorbidity Index (CCI) score is a system used to predict the risk of mortality for patients with multiple comorbidities. It's calculated by summing the weights assigned to different health conditions a patient has.
  The index includes 19 conditions, such as myocardial infarction, congestive heart failure, and cancer, and each is assigned a score based on its predicted impact on mortality. A higher score indicates a higher predicted risk of mortality and lower predicted survival. A score of 0 suggests no significant comorbidities. Scores can range from 0 to 24.
  units on a scale | 3 (2) | 3 (2) | 3 (2) | 3 (4) | 3 (2)

OUTCOME MEASURES:

1. Secondary Outcome: Change in Diabetes Distress (Pre and Post Intervention) Using the Problem Areas in Diabetes (PAID) Tool
Description: Validated tool measuring diabetes distress. Lower score indicates lower diabetes distress (better outcome). 20 item questionnaire, scale 0-100. Scores ≥40 indicate risk of emotional burnout.
  To calculate the change between baseline and follow up (4 months) we calculated the value at follow up minus baseline score.
Time Frame: Measured at baseline and 3-4 months after intervention
Population: Four participants were not included in the final analysis due to protocol deviations: three attended Insulin safe start[29] structured education during the trial to meet their medical needs, one of whom was of mixed ethnicity, and another completed 100% DSME instead of the randomised 60%. A further 3 were lost to follow up
Measure: Mean (Standard Error); unit: adjusted change score -dif in pre & post
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 30 | 27 | 28 | 28
adjusted change score -dif in pre & post | 8.14 (2.44) | 7.14 (2.53) | 2.54 (2.52) | -6.5 (2.48)

2. Secondary Outcome: • Mental Health Quality of Life Outcome Measures (Pre and Post Intervention) Using the PROMIS-Global Health V1.2 Scale
Description: Validated tool measuring health related quality of life. The PROMIS Global-10 is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
  T-score <50 worse than average, >50 better than average.
  To calculate the change between baseline and follow up (4 months) we calculated the value at follow up minus baseline score.
Time Frame: Measured at baseline and 3-4 months after intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change score -dif in pre & post
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 30 | 27 | 28 | 28
change score -dif in pre & post | 3.0 (6.18) | 1.07 (4.77) | -.88 (7.67) | -.61 (8.22)

3. Secondary Outcome: Physical Health Quality of Life Outcome Measures (Pre and Post Intervention) Using the PROMIS-Global Health V1.2 Scale
Description: as for outcome 2
Time Frame: 3-4 months post baseline
Population: Mental health Quality of life outcome measures (pre and post intervention) using the PROMIS-Global Health V1.2 scale
Measure: Mean (Standard Deviation); unit: change score -dif in pre & post
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 30 | 27 | 28 | 28
change score -dif in pre & post | 2.27 (6.95) | 2.58 (4.92) | -.67 (6.56) | .48 (7.15)

4. Primary Outcome: Change in DSMQ Diabetes Self Management Questionnaire Measuring Diabetes Self Management Skills Pre and Post Intervention
Description: Diabetes self management questionnaire with good interrater reliability. Higher score indicates better self management. 20 item questionnaire, scale 0-10 with some items reversed scored. Total score added together and then divided by 60. Scores can range form 0-10. A higher score indicates better self management.
  To calculate the change between baseline and follow up (4 months) we calculated the value at follow up minus baseline score.
Time Frame: 3-4 months post baseline
Population: 3 lost to follow up, 4 removed as not per protocol
Measure: Median (Standard Deviation); unit: change score (difference in pre-post)
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 30 | 27 | 28 | 28
change score (difference in pre-post) | .96 (2.75) | 1.08 (2.0) | .28 (1.24) | -.17 (1.38)

ADVERSE EVENTS:
Time Frame: from enrolment until end of follow-up, up to 20 weeks
Description: all adverse events reported as per protocol
Groups:
- Group 1: 3 participants had adverse events none study related - hospitalisation for exacerbations of existing health conditions.
- Group 2; Group 3: 0 adverse events
- Group 4: 1 participant had adverse event none study related - hospitalisation for exacerbations of existing health conditions.
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/27 | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 3/30 | 0/27 | 0/28 | 1/28
Other Adverse Events (participants affected / at risk) | 0/30 | 0/27 | 0/28 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=30) | Group 2 (N=27) | Group 3 (N=28) | Group 4 (N=28)
None was deemed to be study related and all were exacerbations of existing health conditions. (General disorders) | 3 (7) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Recruitment from primary care was less effective than anticipated due to challenges in contacting eligible patients and low interest in DSME, consistent with national trends. While recruitment through specialty clinics was more successful, this approach alone lacks scalability for larger trials. Although overall retention and attendance were high, the study sample was predominantly white British, limiting the generalisability of findings to more diverse populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT06419907/Prot_SAP_000.pdf